CLINICAL TRIAL: NCT04432545
Title: Infusion of Allogeneic Stromal Mesenchymal Stem Cells From Wharton´s Jelly in Patients With Diffuse Cutaneous Systemic Sclerosis With Refractory Pulmonary Involvement to Treatment
Brief Title: Infusion of Allogeneic Mesenchymal Stem Cells in Patients With Diffuse Cutaneous Systemic Sclerosis With Refractory Pulmonary Involvement
Status: Available | Type: Expanded Access
Sponsor: Universidad de la Sabana (Other)
Collaborators: Fundación Neumologica Colombiana (Other); Innocell SAS (Industry); Stem Medicina Regenerativa (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-10
Record Dates: First submitted 2020-06-10; First posted 2020-06-16 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Systemic Sclerosis Pulmonary; Pulmonary Hypertension; Pulmonary Fibrosis
Keywords: Refractory systemic sclerosis; systemic sclerosis; pulmonary hypertension; mesenchymal stem cells
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Fibrosis; Scleroderma, Systemic

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Mesenchymal Stem Cells from Wharton ́s jellyintravenous infusion of Mesenchymal Stem Cells from Wharton ́s jelly — Mesenchymal Stem Cells from Wharton ́s jellyintravenous infusion of Mesenchymal Stem Cells from Wharton ́s jelly

SUMMARY:
Progressive SSc is an entity with limited therapeutic alternatives and with asurvival rate of less than 45% in the first 3 to 5 years. The disease causessevere limitation in quality of life ranging from functional limitation to depression. Up to 20% of patients will be refractory to conventional treatment with diseasemodifying anti-rheumatic drugs (DMARDs) and cyclophosphamide therapy.This favors the progression to visceral involvement including gastrointestinal,lung and pulmonary hypertension. The latter being a poor prognostic factor,increases mortality in this group of patients and drastically affects their qualityof life. For this reason, different therapeutic options have been considered including cell transplantation and Stem Cell use. Among the options that have been studied so far are stromal mesenchymal cells from Wharton ́s jelly. These have been used in intravenous infusion or direct application in different disease scenarios ranging from vascular involvement to interstitial lung involvement and cases of pulmonary hypertension, with promising results in terms of clinical progression,improvement in quality of life and prognostic indices. This therapy has proven to have a significant margin of safety at the time of administration and a low rate of adverse events, a self-limiting fever as the most frequent event. Based on the above and considering the possibility of offering patients without therapeutic alternatives to their disease in addition to palliative options, an intravenous infusion of stromal mesenchymal stem cells from Wharton ́s jellyis proposed for three patients with progressive SSc refractory to conventional therapy with pulmonary involvement due to pulmonary hypertension.

Under this premise the question posed in our work is; What are the effects of the infusion of allogeneic mesenchymal stromal cells from Wharton ́s jellyin patients with systemic sclerosis refractory to conventional treatment with Methotrexate or Cyclophosphamide in a population of three patients with severe pulmonary involvement due to pulmonary hypertension.

DETAILED DESCRIPTION:
This study aims to evaluate the therapeutic effects of allogeneic mesenchymal stromal cell infusion as a treatment in patients with systemic sclerosis refractoryto conventional therapy. The group of patients will be collected from the database of families of Stem Regenerative Medicine according to the inclusion and exclusion criteria and verified in the academic committee.

The administration will be intravenously, with a concentration of 2 X 10^6 mesenchymal cells per kilogram of patient weight. The infusions will be carried out nested at cyclophosphamide application cycles ten days after each application of the cyclophosphamide schedule for each patient. To assess safety and therapeutic effects, the occurrence of any adverse event will be described from start of infusion until the conclusion of the trial in six months.

To assess the response, a pre-infusion and sixth-month post-infusion instrument will be applied that includes clinical variables, paraclinical and hemodynamic tests to evaluate skin involvement using the modified RODNAN score, changes in nail capillaroscopy, lung function and structural involvement by high-resolution chest tomography (hrCT), diffusion capacity for carbon monoxide (DLCO) and a 6-minute walk. As part of the cardiovascular assessment, cerebral natriuretic peptide (BNP), transthoracic echocardiogramwill be performed; The Cambridge Pulmonary Hypertension Outcome Review(CAMPHOR) and Sysq will be used as tools for the assessment of pulmonary hypertension. A comparison of these tests before initiation of therapy and after completion of 24 weeks of infusion scheme should be performed.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years and <65 years.• Established diagnosis of systemic sclerosis according to the criteria of theAmerican College of Rheumatology• SSc of poor prognosis, involving life-threatening severe visceralinvolvement (cardiac or pulmonary hypertension ), lack of response toconventional immunosuppressive therapy used in severe forms of thedisease according to the European recommendations of EUSTAR and EBMT, relying on high doses of IV cyclophosphamide (either in monthlybolus for at least six months); or SSc with life-threatening pulmonaryhypertension. Patients may or may not have pulmonary fibrosis.• Signed informed consent.• Presence of a consenting MSC donor• Affiliation to social security

Exclusion Criteria:

* Pregnancy or absence of appropriate contraception throughout the study.• Pulmonary artery systolic pressure (PASP) >75mmHg (onechocardiography or after right heart catheterization);- Theorical DLCO <30%• Calculated creatinine clearance <30 ml/mn/m2• Clinical sign of a congestive heart failure refractory ;• Left ventricular ejection fraction <35% at myocardial scintigraphy orechocardiography;• Chronic atrial fibrillation requiring oral anticoagulant therapy;• Uncontrolled ventricular arrhythmia;• Pericardial effusion with hemodynamic compromise assessed byechocardiography.• Hepatic impairment defined as a persistent increase in transaminases orbilirubin to 3 times normal.• Psychiatric disorders, including drug taking and alcohol abuse.• Active neoplasia or concomitant myelodysplasia, antecedent of neoplasia.• Bone marrow failure defined by neutropenia <0.5 x 109 / L,thrombocytopenia <50 x 109 / L, anemia <8 g / dL, CD4 lymphopenia <200x 106 / L.• Uncontrolled systemic hypertension.• Uncontrolled acute or chronic infection, HIV1, 2 or HTLV-1, 2seropositivity.• Chronic hepatitis B or C active.• Significant exposure to bleomycin, toxic oils, vinyl chloride,trichloroethylene or silica; eosinophilia-myalgia syndrome, eosinophiliafasciitis.• Risk of poor patient compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: John Londono, MD,PhD, Principal Investigator — Universidad de la Sabana
Locations (1):
- Universidad de la Sabana, Chía, Chia, Colombia

REFERENCES:
- [Background] Jaeger VK, Wirz EG, Allanore Y, Rossbach P, Riemekasten G, Hachulla E, Distler O, Airo P, Carreira PE, Balbir Gurman A, Tikly M, Vettori S, Damjanov N, Muller-Ladner U, Distler JH, Li M, Walker UA; EUSTAR co-authors. Incidences and Risk Factors of Organ Manifestations in the Early Course of Systemic Sclerosis: A Longitudinal EUSTAR Study. PLoS One. 2016 Oct 5;11(10):e0163894. doi: 10.1371/journal.pone.0163894. eCollection 2016. PMID 27706206
- [Background] McNearney TA, Reveille JD, Fischbach M, Friedman AW, Lisse JR, Goel N, Tan FK, Zhou X, Ahn C, Feghali-Bostwick CA, Fritzler M, Arnett FC, Mayes MD. Pulmonary involvement in systemic sclerosis: associations with genetic, serologic, sociodemographic, and behavioral factors. Arthritis Rheum. 2007 Mar 15;57(2):318-26. doi: 10.1002/art.22532. PMID 17330281
- [Background] Sullivan KM, Goldmuntz EA, Keyes-Elstein L, McSweeney PA, Pinckney A, Welch B, Mayes MD, Nash RA, Crofford LJ, Eggleston B, Castina S, Griffith LM, Goldstein JS, Wallace D, Craciunescu O, Khanna D, Folz RJ, Goldin J, St Clair EW, Seibold JR, Phillips K, Mineishi S, Simms RW, Ballen K, Wener MH, Georges GE, Heimfeld S, Hosing C, Forman S, Kafaja S, Silver RM, Griffing L, Storek J, LeClercq S, Brasington R, Csuka ME, Bredeson C, Keever-Taylor C, Domsic RT, Kahaleh MB, Medsger T, Furst DE; SCOT Study Investigators. Myeloablative Autologous Stem-Cell Transplantation for Severe Scleroderma. N Engl J Med. 2018 Jan 4;378(1):35-47. doi: 10.1056/nejmoa1703327. PMID 29298160
- [Background] van Laar JM, Farge D, Sont JK, Naraghi K, Marjanovic Z, Larghero J, Schuerwegh AJ, Marijt EW, Vonk MC, Schattenberg AV, Matucci-Cerinic M, Voskuyl AE, van de Loosdrecht AA, Daikeler T, Kotter I, Schmalzing M, Martin T, Lioure B, Weiner SM, Kreuter A, Deligny C, Durand JM, Emery P, Machold KP, Sarrot-Reynauld F, Warnatz K, Adoue DF, Constans J, Tony HP, Del Papa N, Fassas A, Himsel A, Launay D, Lo Monaco A, Philippe P, Quere I, Rich E, Westhovens R, Griffiths B, Saccardi R, van den Hoogen FH, Fibbe WE, Socie G, Gratwohl A, Tyndall A; EBMT/EULAR Scleroderma Study Group. Autologous hematopoietic stem cell transplantation vs intravenous pulse cyclophosphamide in diffuse cutaneous systemic sclerosis: a randomized clinical trial. JAMA. 2014 Jun 25;311(24):2490-8. doi: 10.1001/jama.2014.6368. PMID 25058083